CLINICAL TRIAL: NCT01576601
Title: The Management of Postoperative Craniotomy Pain in Pediatric Patients: A Prospective Cohort Study
Brief Title: The Management of Postoperative Craniotomy Pain in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00051171
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Post Craniotomy Surgery; Cancer; Epilepsy; Vascular Malformations; Craniofacial Reconstructive Surgery
Keywords: pediatrics; acute pain; neurosurgery; Pediatric patients (0-18); postoperative management
MeSH Terms: conditions — Neoplasms; Epilepsy; Vascular Malformations; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hopkins: Pediatric patients (0-18 yo) who are scheduled for craniotomy surgery under general anesthesia. This will include patients undergoing brain surgery for cancer, epilepsy, vascular malformations, and craniofacial reconstructive surgery. Patients will receive routine postoperative management and treated for pain based on institutional routine. We will follow patients for the first 5 post-operative days or until discharge, whichever comes first.
- Childrens Hospital of Philadelphia: Pediatric patients (0-18 yo) who are scheduled for craniotomy surgery under general anesthesia. This will include patients undergoing brain surgery for cancer, epilepsy, vascular malformations, and craniofacial reconstructive surgery. Patients will receive routine postoperative management and treated for pain based on institutional routine. We will follow patients for the first 5 post-operative days or until discharge, whichever comes first.
- Childrens Hospital Boston: Pediatric patients (0-18 yo) who are scheduled for craniotomy surgery under general anesthesia. This will include patients undergoing brain surgery for cancer, epilepsy, vascular malformations, and craniofacial reconstructive surgery. Patients will receive routine postoperative management and treated for pain based on institutional routine. We will follow patients for the first 5 post-operative days or until discharge, whichever comes first.

SUMMARY:
The purpose of this prospective, clinical observational trial is to assess the incidence of pain (and analgesia), methods of pain assessment (and by whom), prescribed analgesics, methods of analgesic delivery, and patient/parent satisfaction in patients undergoing craniotomy surgery at three major children's hospitals (Boston Children's Hospital, Children's Hospital of Philadelphia, The Children's Center Johns Hopkins Hospital) in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 0-18 years, who are scheduled to undergo craniotomy surgery for any reason (e.g., brain tumor, epilepsy surgery, craniofacial reconstruction) at either the Boston Children's Hospital, the Children's Hospital of Philadelphia, or the Children's Center of the Johns Hopkins Hospital will be eligible for enrollment.

Exclusion Criteria:

* Patients who remain intubated after surgery. Additionally, we will exclude patients who are allergic to opioids or who have a history of substance abuse

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 200 patients who are scheduled for craniotomy surgery under general anesthesia at 3 major children's hospitals will be eligible. Potential patients include those undergoing brain surgery for cancer, epilepsy, vascular malformations, and craniofacial reconstructive surgery. Following surgery, patients will receive routine postoperative management and treated for pain based on institutional routine. We will follow patients for the first 5 post-operative days or until discharge, whichever comes first.
  Once daily, a study investigator will make an independent pain assessment using an age appropriate, validated tool (FLACC, Pain Face Scale-Revised, self report on a 0-10 scale). The study investigator will also assess overall quality of life and patient/parent satisfaction using a subset of the NRC Picker satisfaction tool and in adolescents a modified QoR-40 (see below).
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
pain assessment | 2 years
  To determine the severity of pain and the compliance of physicians and nurses in implementation of institutionally mandated pain assessment tools by chart review. We will also assess which pain assessment tools are in use by health care providers in the 3 participating institutions along with compliance with frequency of pain assessment based on institutional policy.

SECONDARY OUTCOMES:
patient/parent satisfaction | 2 years
  To independently determine patient/parent satisfaction and quality of recovery (QOR). Daily, an investigator will use a validated, standardized parental satisfaction tool (a subset of the NRC Picker satisfaction tool) and in adolescents a modified QoR-40.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Morad A, Winters B, Stevens R, White E, Weingart J, Yaster M, Gottschalk A. The efficacy of intravenous patient-controlled analgesia after intracranial surgery of the posterior fossa: a prospective, randomized controlled trial. Anesth Analg. 2012 Feb;114(2):416-23. doi: 10.1213/ANE.0b013e31823f0c5a. Epub 2011 Dec 9. PMID 22156333
- [Background] Morad AH, Winters BD, Yaster M, Stevens RD, White ED, Thompson RE, Weingart JD, Gottschalk A. Efficacy of intravenous patient-controlled analgesia after supratentorial intracranial surgery: a prospective randomized controlled trial. Clinical article. J Neurosurg. 2009 Aug;111(2):343-50. doi: 10.3171/2008.11.JNS08797. PMID 19249923
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Derived] Maxwell LG, Buckley GM, Kudchadkar SR, Ely E, Stebbins EL, Dube C, Morad A, Jastaniah EA, Sethna NF, Yaster M. Pain management following major intracranial surgery in pediatric patients: a prospective cohort study in three academic children's hospitals. Paediatr Anaesth. 2014 Nov;24(11):1132-40. doi: 10.1111/pan.12489. Epub 2014 Jul 29. PMID 25069627